CLINICAL TRIAL: NCT03959007
Title: Impact of Supportive Care on the Experience of Hospitalization of Patients Staying in the Protected Area of the Department of Blood Diseases
Acronym: ASTERIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017_43; 2017-A03453-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-04-10; First posted 2019-05-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Acute Leukemia; Hematopoietic Stem Cell Transplantation (SCT); Aplasia
Keywords: Aesthetic care; Transplant; Well-being; Anxiety; Supportive care
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Usual therapy and complete 3 questionnaire at 3 times during hospitalization : Spielberger State-trait Anxiety Inventory + FACT-Leu quality of life and well-being OMS status
  Interventions: Other: Questionnaire
- Experimental (Experimental): 9 consultations (3 x 3 sessions during hospitalization) of aesthetic care will be provided to patient include in experimental arm and 3 times questionnaires (Spielberger State-trait Anxiety Inventory + FACT-Leu quality of life and well-being OMS status)
  Interventions: Other: Aesthetic therapy sessions; Other: Questionnaire

INTERVENTIONS:
Other: Aesthetic therapy sessions — Only for experimental arm at 3 times during hospitalization
  Arms: Experimental
Other: Questionnaire — Both arm at 3 times during hospitalization

SUMMARY:
Patients with acute leukemia or received SCT are hospitalized in protected area, at least for 28 days. In this area, there is some rules like: controlled-visit, protective-clothing….so patient are in social and familial isolation condition.

During their hospitalization, patients are confront to aggressive treatment and psychological distress related to potentially death.

Emergency hospitalization, illness, controlled environment, aggressive treatment and potential complications place patients in a context of anxiety-provoking.

Aesthetic therapy is a new supportive care in cancer therapy access on improving well-being, relaxation and body image.

This supportive care is already used in cancerology department, particularly in breast cancer patients.

In our department, a few patient received aesthetic care during their hospitalization and they appreciated these sessions and impact on well-being was immediately.

Moreover only 6 sessions was proposed and effect on anxiety wasn't measurable Aesthetic care improve well-being but impact on anxiety is unknown. In this study we evaluate the impact off socio aesthetic on the quality off life and anxiety. We evaluate this impact by 3 questionnaires at 3 times during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patient (male or female) ≥18 years old
* Hospitalized patient in restricted area than 21 days
* Patient with acute leukemia (induction or relapse)
* Patient hospitalized for hematopoietic stem cell transplantation
* Written Inform consent must be obtained before inclusion and randomization
* Patient affiliated to and covered by social security for standard care

Exclusion Criteria:

* Patient hospitalized for another disease
* Inability to receive study information and/or understand/speak French
* Inability to give informed consent
* Legal incapacity (people in jail) or under supervision (i.e. guardianship or curatorship)
* Already include in this study on a previous hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
Anxiety score by Spielberger questionary | Baseline and Aplasia (between day10 and 14 of hopitalization)
  Difference between the 2 Arms on anxiety score (Spielberger questionary: composed of 20 items rated from 1 to 4 points)

SECONDARY OUTCOMES:
Anxiety score by Spielberger questionary | Baseline and day 21 of hospitalization
  Difference between the 2 Arms on anxiety score (Spielberger questionary: composed of 20 items rated from 1 to 4 points)
Quality of Life Assessment using the Functional Assessment of Cancer Therapy-Leukemia (FACT-LEU). | Baseline, Aplasia and day 21 of hospitalization
  Difference betwenn the 2 Arms on quality of life score FACT-LEU questionnary: Leukemia Subscale (LeuS): Range:0-68. To derive: Subtract the answers from "4" for each of the 17 questions, Range: 0-176.
Well-being score | Baseline, Aplasia and day 21 of hospitalization
  Difference between the 2 Arms on well-being score (OMS questionary)

CONTACTS AND LOCATIONS:
Overall Officials: Celine Berthon, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, France